CLINICAL TRIAL: NCT00873314
Title: Bed Rest for Arrested Threatened Preterm Labor. Pilot Study for the Design of a Randomized Controlled Clinical Trial.
Brief Title: Bed Rest for Threatened Preterm Labor. Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Collaborators: Unidad de Investigación Clínica y Epidemiológica Montevideo (Other)
Responsible Party: Fernando Althabe, Institute for Clinical Effectiveness and Health Policy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIHR01-2003
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Bedrest; Premature Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bed rest (Experimental)
  Interventions: Behavioral: Bed rest
- Activity restriction (Placebo Comparator)
  Interventions: Behavioral: Activity restriction

INTERVENTIONS:
Behavioral: Bed rest — The woman assigned to the bed rest group, will be instructed to keep in bed for the study period of four days and will be allowed to go to the toilet
  Arms: Bed rest
Behavioral: Activity restriction — Women assigned to activity restriction group will do the restriction of activities during four days.During the activity restriction phase the women will be allowed to ambulate at home, work at home (home office), child care, household tasks, meal preparation or any forceless activities.
  Arms: Activity restriction

SUMMARY:
The aim of the pilot trial is to assess at what extend women with arrested threatened preterm labor change their activity patterns at home in response to bed rest prescription.

An area of concern for the design of a trial is the strength of health provider's recommendation to change women's behaviors, and their compliance with bed rest recommendations. The study was a randomized parallel design. The intervention group consisted of total bed rest for four days (with allowance to go to the toilet). The control group consisted in the restriction of activities during four days.

ELIGIBILITY:
Inclusion Criteria:

* Every woman admitted to hospital during the antenatal period because of an episode of TPL. If the attending physician decides that the woman is ready for hospital discharge the woman will be eligible for the study.

Exclusion criteria:

* Multiple pregnancy
* Premature rupture of membranes
* Cervical cerclage and whenever the attendant physician considers that the woman is not eligible to be randomized to bed rest or activity restriction.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The outcome was the amount of activity. In order to measure the outcome, we used: a) an accelerometer which was delivered to the woman at home and b) a diary record that the woman fulfilled during the study. | Four days

CONTACTS AND LOCATIONS:
Locations (1):
- Pereira Rossell Hospital, Montevideo, Uruguay

REFERENCES:
- See also: Institute for Clinical Effectiveness and Health Policy — http://www.iecs.org.ar/
- See also: School of Medicine of the University of the Republic — http://www.fmed.edu.uy/
- See also: Clinical and Epidemiological Research Unit Montevideo — http://www.unicem-web.org/